CLINICAL TRIAL: NCT02891031
Title: The Effects of Rhus Coriaria L. on Serum Uric Acid Levels
Acronym: SomaghUricA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of Internal medicine and Endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11541-01-01-95
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Hyperuricemia
Keywords: Rhus; Medicine, Traditional; Herbal medicine; Uric acid
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhus (Somagh) (Active Comparator): 500 mg twice daily after meal for 6 weeks
  Interventions: Drug: Rhus (Somagh)
- Placebo (Placebo Comparator): 500 mg twice daily after meal for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rhus (Somagh) — 500 mg twice daily after meal for 6 weeks
  Other Names: Somagh
  Arms: Rhus (Somagh)
Drug: Placebo — 500 mg twice daily after meal for 6 weeks
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effects of Rhus coriaria L. (Rhus) commonly known as "Somagh" on serum uric acid levels.

DETAILED DESCRIPTION:
Rhus coriaria L.(Rhus) is a well-known spice widely consumed in the world which has also been utilized extensively for medicinal purposes. The antioxidant components of this plant made it a favorable target for laboratory and animal studies in different conditions such as oxidative stress cytotoxicity, diabetes and hyperlipidemia. Rhus (Somagh) is found in temperate and tropical regions worldwide, often growing in areas of marginal agricultural capacity. Rhus is used as an herbal remedy in traditional medicine because of its assumed analgesic, antidiarrheic, antiseptic, anorexic and antihyperglycemic properties. The fruits of Rhus contain flavonols, phenolic acids, hydrolysable tannins, anthocyans and organic acids such as malice, citric and tartaric acids. Some studies have shown that polyphenols could have beneficial effects on cardiovascular disease and cancer and could be regarded as bioactive compounds with a high potential health-promoting capacity. Phenolic compounds inhibit lipid peroxidation, scavenge the superoxide anion and hydroxyl radical, and enhance the activities of detoxifying enzymes.

Uric acid (UA; 7,9-dihydro-1H-purine-2,6,8(3H)-trione) has been implicated as a risk factor and cause of numerous disease states. Some disease states, such as gout, hypertension, and cardiovascular disease, have been shown to result when UA levels in the blood are too high. Hyperuricemia predicts the development of hypertension in the general population, and an independent positive correlation between UA levels and the occurrence of hypertension has been reported. Hyperuricemia may also be a risk factor for cardiovascular disease, myocardial infarction, and stroke.

The manipulation of serum UA levels has become a popular strategy in the treatment of a variety of diseases. This is either accomplished through dietary and lifestyle changes or through treatment with UA reducing drugs.

The aim of this study is to evaluate the effects of Rhus coriaria L. (Rhus) commonly known as Somagh on serum uric acid levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Serum uric acid levels that need medical treatment
* Gout
* Diabetes mellitus
* Hypo. or hyperthyroidism
* Any systemic illnesses e.g. liver cirrhosis, acute or chronic renal failure, heart failure
* Use of drugs: Uric acid lowering agents
* Pregnancy
* Lactation
* History of allergic reaction to Somagh

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
serum uric acid levels | 6 weeks

SECONDARY OUTCOMES:
Number of patients with adverse events. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gholamhossein Ranjbar Omrani, MD, Principal Investigator — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences; Seiyed Mohammad Hosseini-Saadi, MD, Principal Investigator — Department of Internal Medicine, Shiraz University of Medical Sciences
Locations (1):
- Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No